CLINICAL TRIAL: NCT00761800
Title: Study for Dermatological Evaluation of Topic Compatibility (Primary and Accumulated Dermal Irritability, Dermal Sensitivity) of Dermacyd Teen Care Tangerina Mix .
Brief Title: Dermacyd Teen Care Tangerina Mix - Compatibility
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study director, Sanofi-aventis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: LACAC_L_04087
Record Dates: First submitted 2008-09-29; First posted 2008-09-30 (Estimated); Last update posted 2009-05-29 (Estimated); Status verified 2009-05

CONDITIONS: Hygiene
MeSH Terms: interventions — Lactic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Lactic acid

SUMMARY:
The purpose of this study is to demonstrate the absence of irritation potential (primary dermal irritability and cumulated dermal irritability) and allergy (sensibilization) of the product Dermacyd Teen Care Tangerina Mix.

ELIGIBILITY:
Inclusion Criteria:

* Phototype Skin I,II, III e IV
* Integral skin test in the region

Exclusion Criteria:

* Lactation or gestation
* Use of Anti-inflammatory and/or immuno-Supression drugs 1 month before the study
* Personal history of atopy
* History of sensitivity or irritation for topic products
* Active cutaneous disease
* Use of new drugs or cosmetics during the study

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2008-05; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
The absence of primary and accumulated dermal irritability will be evaluated using International Contact Dermatitis Research Group (ICDRG) scale. | Throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Jaderson Lima, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, São Paulo, Brazil